CLINICAL TRIAL: NCT05971524
Title: Effect of 4 Weeks of Oral 6-bromotryptophan on Safety, Pharmacokinetics and Efficacy in Metabolic Syndrome Individuals (2022)
Brief Title: Effect of Oral 6-bromotryptophan on Safety, Pharmacokinetics and Efficacy in Metabolic Syndrome Individuals
Acronym: BROMO
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nordin Hanssen (Other)
Responsible Party: Sponsor-Investigator, Nordin Hanssen, Principal Investigator, Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL83061.018.22
Record Dates: First submitted 2023-04-20; First posted 2023-08-02 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Metabolic Syndrome; Diabetes Mellitus
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: A phase I/II, dose finding, placebo controlled, double blinded trial
Who Masked: Participant, Investigator
Masking Description: To maintain the blinding of the subject and investigators, the identifying labels will be removed from the intervention product at the AMC pharmacy. The study product will be labelled with subject specific information prior to delivery to the study physician, who will hand over the intervention to the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): An oral placebo capsule once daily for 4 weeks
  Interventions: Dietary Supplement: Placebo
- 2mg 6-BT (Experimental): 2 mg of 6-BT as an oral capsule once daily for 4 weeks
  Interventions: Dietary Supplement: 6-BT
- 4mg 6-BT (Experimental): 4 mg of 6-BT as an oral capsule once daily for 4 weeks
  Interventions: Dietary Supplement: 6-BT
- 8mg 6-BT (Experimental): 8 mg of 6-BT as an oral capsule once daily for 4 weeks
  Interventions: Dietary Supplement: 6-BT

INTERVENTIONS:
Dietary Supplement: 6-BT — 2,4 or 8mg of 6-BT once daily for 4 weeks
  Arms: 2mg 6-BT; 4mg 6-BT; 8mg 6-BT
Dietary Supplement: Placebo — A placebo capsule once daily for 4 weeks
  Arms: Placebo

SUMMARY:
Safety, pharmacokinetics and efficacy of a novel endogenous plasma metabolite, 6-bromotryptophan, will be established in metabolic syndrome/ insulin resistant participants.

DETAILED DESCRIPTION:
Rationale:

A newly identified endogenous plasma microbiome-derived tryptophan metabolite, 6-bromotryptophan (6-BT), was associated with preserved beta-cell function and diminished circulating T cell count in (T1D) type 1 diabetes patients. Anti-inflammatory and insulin-secratogogue effects were established in in vitro- and murine studies in both the setting of type 1 and type 2 diabetes. Also, 6-BT did not show any toxic effects in cells or in vivo experiments. In order to obtain safety data before the investigators progress to an efficacy study in T1D, the investigators aim to perform a phase I/II trial of 6-BT in metabolic syndrome individuals. If safe, 6-BT may hold a promise as a food supplement in type 1 and 2 diabetes.

Objective: To assess safety, pharmacokinetics and efficacy of oral dosage of 6-BT in individuals with metabolic syndrome Study design: A phase I/II, dose finding, placebo controlled, double blinded trial.

Study population: Metabolic syndrome individuals or participants with insulin resistance, age 35-70 years, without use of medication.

Intervention (if applicable): Participants will be given placebo, 2mg, 4mg or 8mg of 6-BT capsules once daily for 4 weeks (n=9 per arm, total of 36 participants).

Main study parameters/endpoints:

The principal outcome will be patient safety and tolerability (biochemical parameters of kidney and liver function and complete blood count, adverse events) in relation to improvements in glucose homeostasis (mixed-meal tests and continuous glucose monitoring). Secondary read-outs will include changes in: immunological profile (ex vivo stimulation of monocytes, and immunophenotyping of peripheral blood mononuclear cells (PBMC)) and gut microbiome composition (16s ribosomal ribonucleic acid (rRNA) sequencing). Also, liver fat content will be determined before and at end of the trial by MRI. As this food derived metabolite is given to humans for the first time, the investigators will also study its pharmacokinetics by measuring serum 6-BT concentrations in serum and urine at different time-points after oral intake.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

6-BT is an endogenous (food tryptophan derived) metabolite found in the human circulation. Our previous trail has shown that fecal microbiota transplantations (FMT) can modulate and increase plasma 6-BT levels with a positive association with C-peptide (as marker of pancreatic beta cells function). Additionally, recent investigations have linked higher plasma 6-BT levels with lower risk of kidney disease progression, supporting the health benefits of 6-BT beyond T1D. Hence, the investigators do not foresee major adverse reactions. As there is an urgent need for halting diabetes progression, patients would benefit from the development of new endogenously occurring therapeutic agents.

ELIGIBILITY:
Inclusion Criteria:

• Metabolic syndrome, defined as:

- ≥3 criteria out of the 5 following criteria:

* fasting plasma glucose ≥5.6 mmol/L
* triglycerides ≥1.7 mmol/L
* waist circumference ≥102 cm
* high-density lipoprotein cholesterol ≤1.04 mmol/
* blood pressure ≥130/85 mm Hg.

AND/ OR Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) (>2.5)

* Male
* Caucasian
* 35-70 years old

Exclusion Criteria:

* Use of systemic medication (except for paracetamol), including proton pump inhibitors, antibiotics and pro-/prebiotics in the past three months or during the study period.
* A history of a cardiovascular event
* A history of cholecystectomy
* Overt untreated gastrointestinal disease or abnormal bowel habits
* Liver enzymes>2.5 fold higher than the upper limit of normal range
* Smoking
* Exclusion criterion for MRI liver (see E4_BROMO_vragenlijst MRI)
* Alcohol abuse

Ages: 35 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 4 weeks
  Number of adverse events
renal function | 4 weeks
  Number of participants with a decreased kidney function, defined as a rise in serum creatinine of >26,5 micromol/L in 48 h
Questionnaires | 4 weeks
  Changes in Gastro-intestinal Quality of Life Index (GIQLI score) (points). The minimum and maximum score are 31 and 155 points respectively, and a higher score reflects a better outcome.
Occurence of anemia | 4 weeks
  Number of patients with Hb < 8,5 mmol/L
Changes in leucocytes | 4 weeks
  Number of patients with leucocytes <4,0 or >10,5 x10E9 cells/L
Changes in trombocytes | 4 weeks
  Number of patients with trombocytes <150 x 10E9 cells/L
Changes in aspartate aminotransferase (AST) | 4 weeks
  Number of patients with AST > 43 IU/L
Changes in alanine aminotransferas (ALT) | 4 weeks
  Number of patients with ALT > 45 IU/L
Changes in alkaline phosphatase (ALP) | 4 weeks
  Number of patients with ALP > 126 IU/L
Changes in Gamma-glutamyltransferase (GGT) | 4 weeks
  Number of patients with GGT > 117 IU/L
Changes in total bilirubin | 4 weeks
  Number of patients with total bilirubin > 24 micromol/L
Mixed meal test | 4 weeks
  Changes in area under the curve (AUC) of glucose after mixed-meal test
Mixed meal test | 4 weeks
  Changes in area under the curve (AUC) of insulin after mixed-meal test
Time-in-range | 4 weeks
  Increase in Time-in-range (TIR,%), a parameter of continuous glucose monitoring devices, where TIR can be between 0 and 100%. A higher TIR reflects a better outcome.
Continuous glucose monitoring | 4 weeks
  Decrease in glucose variability (GV, %), a parameter of continuous glucose monitoring devices, where GV can be between 0 and 100%. A lower GV reflects a better outcome.
Glycemic control | 4 weeks
  Changes in fasting glucose (mmol/L)

SECONDARY OUTCOMES:
Intestinal microbiota composition | 4 weeks
  Changes from baseline of relative abundance (%) of bacterial phyla, genera and species between groups and within participants.
Immunologic profile | 6 weeks
  Absolute counts of different immunologic cell types using Cytometry by time of flight (CyTOF) mass cytometry at baseline, 4 weeks and 6 weeks.
6-BT pharmacokinetics | 6-BT pharmacokinetics as described above will be performed at baseline and after 4 weeks.
  Quantitatively measuring plasma concentrations of 6-BT at -15, 30, 60, 90, 120, 240 and 300 minutes following 6-BT capsule ingestion
Hepatic stiffness | 0 and 4 weeks
  Hepatic stiffness will be determined non-invasively by MRI using a special hepatic scanning protocol of 30 minutes
Hepatic fat content | 0 and 4 weeks
  Hepatic fat content will be determined non-invasively by MRI using a special hepatic scanning protocol of 30 minutes
Dietary intake | 4 weeks
  Participants are asked to fill out an online dietary questionnaire for the 3 days prior to study visit 2,3,4,5 and 7
Low-density lipoprotein (LDL) | 4 weeks
  Changes in LDL (mmol/L)
High-density lipoprotein (HDL) | 4 weeks
  Changes in HDL (mmol/L)
Triglycerides | 4 weeks
  Changes in triglycerides (mmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Nordin MJ Hanssen, dr., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No